CLINICAL TRIAL: NCT07192510
Title: Pancake Oral Immunotherapy For Egg Allergy In Inducing Tolerance (POET)
Brief Title: Pancake Oral Immunotherapy For Egg Allergy In Inducing Tolerance
Acronym: POET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Chong Kok Wee, Principal Investigator, KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB Ref: 2020/3072; PAEDSACP-TCL/2021/RES/002 (Other Grant/Funding Number: Paediatrics Academic Clinical Programme)
Record Dates: First submitted 2025-08-25; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Egg Allergy
Keywords: oral immunotherapy
MeSH Terms: conditions — Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Pancake Oral Immunotherapy
  Interventions: Other: Pancake oral immunotherapy
- Control (No Intervention): Standard of care - strict egg avoidance

INTERVENTIONS:
Other: Pancake oral immunotherapy — The baked egg tolerant group underwent a 4-dose initial escalation (at intervals of 20-30 minutes) with pancakes in hospital (37.5 mg, 75 mg, 150 mg, 300 mg egg protein) to determine the home starting dose of pancake. The dose tolerated was one which resulted in no more than mild transient (not lasting more than 20 minutes) symptoms (e.g. itchy mouth) - transient Grade 1 symptoms. The home starting dose (taken daily at home) was one step below the tolerated dose, to minimise risk of allergic reactions at home, particularly as the presence of co-factors might decrease reaction threshold. Those reacting at 37.5 mg or 75 mg would not begin OIT with pancakes but instead began with cookies. Updosing visits were performed in the hospital at approximately 4 weekly intervals. Participants were kept at the pancake daily maintenance dose (2500 mg) for a minimum of 16 weeks, or total OIT duration of 18 months, whichever earlier
  Other Names: OIT
  Arms: Active

SUMMARY:
Oral immunotherapy (OIT) using raw/ cooked egg has good desensitisation outcomes but is associated with frequent and sometimes severe adverse events (anaphylaxis is not uncommon). OIT using baked egg is less effective at inducing desensitisation but has a better safety profile. The compliance to daily consumption of baked egg products (muffins/ biscuits) after a negative baked egg challenge in egg allergic patients has also been reported to be poor, secondary to taste fatigue in children and need for frequent baking. A study using baked egg OIT had 38% withdrawal due to difficulties in ingesting the baked egg product daily. Pancakes, traditionally described as a flat cake prepared from a starch-based batter containing egg and milk and cooked on a hot surface for 5-7 minutes, is likely to be less allergenic than cooked egg because of the wheat matrix but more allergenic than baked egg. To date, there are no published studies investigating the use of pancakes in egg OIT. The investigators hypothesize that pancakes are more effective than baked eggs in inducing desensitisation and sustained unresponsiveness while reducing the risk of adverse events associated with egg OIT.

ELIGIBILITY:
Inclusion Criteria:

* Allergic to 4.443g egg protein or less, at baseline egg open food challenge OR Convincing clinical reaction to egg within past 6 months (or failed a clinical egg food challenge in last 6 months) AND evidence of current sensitization (positive SPT or egg-specific IgE performed within the last 3 months)

Exclusion Criteria:

Subjects meeting any of the exclusion criteria at baseline will be excluded from participation.

* Required previous admission to an intensive care unit for management of an allergic reaction.
* Children with a past history of egg allergy currently consuming egg-containing products other than extensively-heated egg in baked foods (e.g. biscuits, cakes).
* Developed severe anaphylaxis to egg or egg-containing products requiring more than 2 adrenaline auto-injectors or intravenous adrenaline infusion.
* Poorly controlled asthma within the previous 3 months (as defined by clinician judgement with reference to the ICON guidelines).
* Moderate-severe eczema despite appropriate use of emollients (eczema is not otherwise an exclusion criteria).
* Clinically significant chronic illness (other than asthma, rhinitis or eczema).
* History of symptoms of eosinophilic oesophagitis, irrespective of cause.
* Undergoing specific immunotherapy to another allergen and within the first year of treatment.
* Receiving anti-IgE therapy, oral immunosuppressants, beta-blocker or ACE inhibitor.
* Pregnancy.
* Unwilling or unable to fulfil study requirements.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving desensitisation - tolerating a cumulative dose of 4443 mg cooked egg protein | 12-18 months

SECONDARY OUTCOMES:
Proportion of participants achieving sustained unresponsiveness - tolerating a cumulative dose of 4443 mg cooked egg protein after 6-8 weeks of egg abstinence | 12-18 months
Number of treatment-related adverse reactions as assessed by CoFAR Grading | 12-18 months
  Consortium for Food Allergy Research (CoFAR) grading system: Grade 1-2 (Mild-moderate reactions), Grade 3-5 (Anaphylaxis)
Change in skin prick test wheal size to egg white | 12-18 months
Change in serum IgE levels to egg white, ovomucoid, ovalbumin | 12-18 months
Change in Food-Allergy Quality of Life Questionnaire (FAQL-Q) scores | 12-18 months
  Total mean score range 0-6. The higher the mean score the poorer the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT07192510/Prot_SAP_000.pdf